CLINICAL TRIAL: NCT06643403
Title: Age-related Changes in Retinal Oxygen Extraction in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc. Prof. Priv.-Doz. Dr.med.univ. PhD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-26052024
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants; Retinal Oxygen Extraction
MeSH Terms: interventions — Oxygen; Gases; Inhalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): SAUERSTOFF medizinisch, Messer GmbH, Industriestrasse 5, 2352 Gumpoldskirchen, Austria Dose: min. 95.5%, breathing for max. 45 minutes
  Interventions: Drug: Oxygen 100% Gas for Inhalation

INTERVENTIONS:
Drug: Oxygen 100% Gas for Inhalation — SAUERSTOFF medizinisch, Messer GmbH, Industriestrasse 5, 2352 Gumpoldskirchen, Austria
  Dose:
  min. 95.5%, breathing for max. 45 minutes

SUMMARY:
It has been found that several systemic and ocular diseases are associated with impaired retinal oxygen extraction. In the present study, retinal oxygen extraction will be measured in different age groups in order to identify age related changes in otherwise healthy subjects. In addition, the study will explore short-term changes in retinal metabolism induced by breathing pure oxygen. Measurements will be performed with dynamic vessel analyzer and laser speckle flowgraphy to evaluate retinal blood flow and retinal oxygen saturation, in order to calculate retinal oxygen extraction.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 80 years
* Signed informed consent
* Normal ophthalmic findings, unless the investigator considers an abnormality to be clinically irrelevant for the purpose of the study
* Normal findings in the medical history, unless the investigator considers an abnormality to be clinically irrelevant for the purpose of the study
* Nonsmokers

Exclusion Criteria:

* Abuse of alcoholic beverages or drugs
* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnant or breast-feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Retinal oxygen extraction in different age groups | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Vienna, Austria